CLINICAL TRIAL: NCT04451759
Title: Exploration by UHF MRI of Hypothalamic Networks Associated to Feeding in Obesity and Anorexia
Acronym: HYPOTHALNET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-45
Record Dates: First submitted 2020-06-22; First posted 2020-06-30 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-06

CONDITIONS: Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- healthy controls (Active Comparator)
  Interventions: Other: MRI exploration
- Anorexia (Experimental)
  Interventions: Other: MRI exploration
- Obesity (Experimental)
  Interventions: Other: MRI exploration

INTERVENTIONS:
Other: MRI exploration — ultra high field (7T) magnetic resonance imaging

SUMMARY:
Food intake is a motivated behaviour that consists of seeking, selecting and ingesting nutritional resources from the environment. Its main function is therefore, depending on these conditions, to ensure the supply, in adequate quantities, of the energy and biochemical substrates necessary for the proper functioning and need of the body. Thus, in addition to maintaining the body's fat mass level stable, dietary behaviour is part of the energy homeostasis system and is thus regulated and maintained by the central nervous system.

Although diet regulation involves several brain regions, the way in which these different regions communicate with each other and influence each other to orchestrate appropriate eating behaviour is not yet fully characterized. Among the structures of this network, the hypothalamus, a small structure (less than 1 cm3 in humans) composed of several nuclei such as the lateral hypothalamus, the arched nucleus or the lateral tuberal nucleus plays a crucial role.

The investigators propose to use ultra high field (7T) magnetic resonance imaging equiping the CEMEREM (CHU Timone, APHM, Marseille) to better characterize the role of this crucial small structure in food intake networks in order to better understand the impact of these structural and functional disorders observed in patients with anorexia nervosa and obesity compared to a control population without eating behaviour disorders.

ELIGIBILITY:
Inclusion Criteria:

* No depression (HADS and BECK scores)
* No contraindication to 7T MRI
* Subject with with social insurance
* Subject who has signed the informed consent

For obese patients

* Body mass index > 30kg/m2
* Body diameter < 60cm (compatible with 7T MR scanner tube)

For anorexic patients

* mental anorexia according to DMS-V
* Body mass index < 17kg/m2

For healthy controls

* 18.5kg/m2<Body mass index < 25kg/m2
* no feeding behavioral disturbance (SCOFF and EAT 26)

Exclusion Criteria:

* Pregnant or parturiente woman
* subject with other neurological or neuropsychiatric diseases
* subject with addiction

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-06-25 (Actual); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
MRI exploration conducted at 7T | 2 years
  Mapping of MRI parameters of 4 sub-regions of the hypothalamus, in order to determine whether the sensitivity of quantitative T1 to 7T imaging at very high resolution can reveal microstructure variations in the 4 sub-regions of the hypothalamus in patients suffering from obesity or anorexia nervosa compared to a control population without eating disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Olivier ARNAUD, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No